CLINICAL TRIAL: NCT05673915
Title: Pilot Study of Transcranial Direct Current Stimulation (tDCS) to Treat Epilepsy
Brief Title: Study of Transcranial Direct Current Stimulation to Treat Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian N. Lundstrom, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-008944
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Focal Epilepsy; Generalized Onset Epilepsy; Sleep-related Epileptic Encephalopathy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- tDCS Treatment A (Low Amplitude) (Experimental): Subjects with focal epilepsy that is not well-controlled on anti-seizure medications will receive 2 different treatments periods, each lasting 2 months, of transcranial direct current stimulation (tDCS). The initial treatment stimulation will be completed during the first 2-months.
  Interventions: Device: ActivaDose II 0.1 mA transcranial direct current stimulation (tDCS)
- tDCS Treatment B (High Amplitude) (Experimental): Subjects with focal epilepsy that is not well-controlled on anti-seizure medications will receive 2 different treatments periods, each lasting 2 months, of transcranial direct current stimulation (tDCS). The last treatment stimulation will be completed during the following 2-months.
  Interventions: Device: ActivaDose II 2.0 mA transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: ActivaDose II 0.1 mA transcranial direct current stimulation (tDCS) — Stimulation setting 0.1 mA daily for a 2-month period. Each daily treatment will last for approximately 30 minutes.
  Arms: tDCS Treatment A (Low Amplitude)
Device: ActivaDose II 2.0 mA transcranial direct current stimulation (tDCS) — Stimulation setting 2.0 mA daily for a 2-month period. A Each daily treatment will last for approximately 30 minutes.
  Arms: tDCS Treatment B (High Amplitude)

SUMMARY:
The purpose of this research is to see to what extent electrical stimulation applied to the scalp (transcranial direct current stimulation or tDCS) can reduce the number and intensity of epileptic seizures.

DETAILED DESCRIPTION:
tDCS for treatment of epilepsy has been studied previously with results suggesting that it can lead to a notable seizure reduction for a limited time period after the cessation of stimulation, e.g., about one month. Here, we assess further aspects of tDCS treatment protocols, including the feasibility and safety of at-home use.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of generalized onset or focal epilepsy or sleep-related epileptic encephalopathy.
* Estimated to have at least 2 countable seizures per month or spike-wave index ≥50%.
* Has not had control with at least 2 anti-seizure medicines.
* Able to maintain a constant medication for duration of the study (rescue meds allowed).
* Subject or legally authorized representative is able to understand consent and keep a seizure diary in English.

Exclusion Criteria:

* A disease likely to progress over course of the study.
* Psychogenic non-epileptic seizures.
* Suicide attempt or psychiatric hospitalization past 2 years.
* A skin condition interfering with scalp electrodes or allergy to silver.
* Women will verify not pregnant, and if applicable, have a serum pregnancy test.
* Implanted devices (e.g. pacemakers)-except VNS, which is allowed.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Seizure Count | 2 months
  Number of seizures experienced by subjects as determined by self-reported seizure diary

SECONDARY OUTCOMES:
EEG interictal discharge frequency | 2 months
  Number of interictal epileptiform discharges observed on electroencephalogram (EEG)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lundstrom, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No